CLINICAL TRIAL: NCT03675113
Title: Effects of Upper Extremity Aerobic Exercise Training on Exercise Capacity and Physical Activity Level in Patients With Chronic Heart Failure
Brief Title: Effect of Upper Extremity Aerobic Exercise Training on Exercise Capacity Patients With Chronic Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was a doctorate thesis and student changed the subject of her thesis.
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, associate professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gazi University 14
Record Dates: First submitted 2018-09-12; First posted 2018-09-18 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Chronic Heart Failure
Keywords: upper extremity aerobic exercise; functional exercise capacity; maximal exercise capacity; respiratory endurance; quality of life; dyspnea; pulmonary function; fatigue; anxiety; depression
MeSH Terms: conditions — Dyspnea; Fatigue; Anxiety Disorders; Depression | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper extremity aerobic group (Experimental): The upper extremity aerobic exercise training with an arm ergometer will be performed in the treatment group so that training intensity will be between 60% and 80% of the maximum heart rate, dyspnea perception will be 3-4 according to Modified Borg Scale and fatigue perception will be 5-6 according to Modified Borg Scale, training duration will be 3 day per a week through 6-weeks.
  Interventions: Other: Upper extremity aerobic exercise
- control group (Sham Comparator): Deep breathing exercises combination with arm movements will be given as a home program in the control group. Training duration will be 3 day per a week through 6-weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Upper extremity aerobic exercise — Range of maximal heart rate will be followed by a polar band during supervised session each week.
  Aerobic exercise will be trained for 30 min-per/day, 3 days/week, 6 weeks. All sessions are being performed by a physiotherapist at cardiopulmonary rehabilitation department.
  Arms: upper extremity aerobic group
Other: Control Group — Deep breathing exercises combinated with arm movements
  Arms: control group

SUMMARY:
Heart failure is a cardiac structural or functional disorder that, despite normal filling pressures, leads to inability to deliver enough oxygen to meet the metabolic needs o tissue. Heart failure is a serious chronic condition that affects a large proportion of the adult population in the world causing high mortality, leading to exercise intolerance and reduced health-related quality of life. Patients included in the cardiac rehabilitation program slow down disease progression, hospitalization decreases, quality of life improves and health expenditures decrease. Despite the frequent use of upper extremities in daily living activities, studies investigating the effect of upper extremity aerobic training on daily living activities, functional exercise capacity and other outcomes are limited. No studies have investigated the effect of upper extremity aerobic exercise training on physical activity level, functional and maximal exercise capacity and other measures in patients with heart failure.

DETAILED DESCRIPTION:
It has been reported that exercise capacity in peak arm exercise is almost 30% lower in heart failure patients. For this reason intolerance to arm exercise is a significant problem in heart failure patients and may contribute to a decrease in performance in activities of daily living. Considering the fact that developments in these patients are caused by vasculature functional adaptation the extremity skeletal muscle and applied limbs, upper extremity exercises may be useful to reduce exercise intolerance during activities requiring continuous arm movement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of chronic heart failure diagnosed at rest below 40% of the left ventricular ejection fraction and class 1-3 according to the New York Heart Association classification
* Optimal medical treatment at least 30 days and clinically stable

Exclusion Criteria:

* Patients with unstable angina pectoris
* Decompensated heart failure
* Primary pulmonary hypertension
* Complex ventricular arrhythmia
* Contraindication to cardiopulmonary exercise testing
* Patients who have had myocardial ischemia in the past 3 months
* Ischemic cerebrovascular events
* Second and third degree atrioventricular block
* Thrombus detected in the left ventricle
* Uncontrolled insulin dependent diabetes mellitus
* Uncontrolled hypertension
* Renal insufficiency
* Acute infection
* Aortic stenosis
* Acute pulmonary embolism
* Mental, musculoskeletal, neurological, or systemic illness that will prevent exercise.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Maximal exercise capacity | Second day
  It will be evaluated using symptom limited cardiopulmonary exercise testing. The cardiopulmonary exercise test will be performed at a progressively increasing speed and grade

SECONDARY OUTCOMES:
Pulmonary function | First day
  Dynamic lung volume measurements will be performed using a spirometry according to the American Thoracic Society and European Respiratory Society criteria.
Respiratory muscle strength | First day
  Maximal inspiratory and expiratory muscle strength will be evaluated a using mouth pressure device.
Pulmonary muscle endurance | First day
  It will be evaluated incremental threshold loading test, in which participants started an initial load of 30% of maximal inspiratory pressure with a 10% increment every 2 minutes.
Peripheral muscle strength | First day
  It will be evaluated using a portable hand held Dynamometer.
Grip strength | First day
  It will be evaluated using a grip dynamometer.
Functional impairment due to dyspnea | First day
  It will be evaluated with modified Medical Research Council Dyspnea Scale (MMRC). MMRC is a baseline assessment of functional impairment attributable to dyspnea from respiratory disease. modiﬁed Medical Research Council (mMRC) Dyspnea Scale, which consist of ﬁve-item scale based on a variety of physical activities that cause a feeling of dyspnea, was used to determine the severity of patients' shortness of breath. The participants read and chose the most appropriate scale option between 0 and 4 that best describes the degree of their pulmonary distress.
Physical activity level | First day
  Physical activity will be evaluated multi sensor activity monitor for 4 consecutive days.
Functional exercise capacity | First day
  Six minute pegboard and ring test (6-PBRT) was applied to assess the functional capacity of the upper limbs. Subjects are asked to move as many rings as possible in 6 minutes, and the score is the number of rings moved during the 6-minute period.
Activity daily of living | Second day
  London Chest Activity Daily of Living Scale is a 15-item scale divided into 4 domains: self-care (4 items), domestic (6 items), physical (2 items), and leisure (3 items).The total score is calculated by summing the domains and ranges from 0 to 75, with higher values indicating more marked limitation in activity daily of living performance.
Quality of sleep | Second day
  Pittsburgh Sleep Quality Index (Turkish version) (PSQI) is a self-reported questionnaire. PSQI evaluates patients' sleep quality. The scale includes 24 questions overall, with 19 questions answered by the person him/ herself and the remaining 5 answered by his/her bed partner or roommate. The first 19 self-answered questions evaluate 7 subscales, subjective sleep quality, sleep latency, duration of sleep, routine sleep activity, sleep disorders, the use of drugs for sleeping, and daytime dysfunction. Each item in the scale is scored between 0 and 3 (no difficulty to severe difficulty). The sum of the 7 subscale scores gives the overall PSQI score. Lower scores show better sleep quality.
Fatigue | Second day
  Fatigue Severity Scale (Turkish version) - Fatigue Severity Scale (FSS) is a self-reported questionnaire. FSS evaluates patient's fatigue severity. This questionnaire includes 9 items and score range for each item from 1 to 7 point (7-point Likert scale). Fatigue Severity Scale score is calculates by deriving an arithmetic mean. Cut-scores of over 4 are indicative of significant fatigue (higher scores show more severe fatigue).
Anxiety and depression | Second day
  Hospital Anxiety and Depression (Turkish version). The test used to determine the risk group of patients in terms of anxiety and depression and consists of 14 questions. Lowest score that patients can get from both subscales is 0, the highest score 21. The cut-off points for the Turkish version of the HAD scale were 10 for the anxiety subscale (HAD-A) and 7 for the depression subscale (HAD-D).
Quality of life scale | Second day
  Minnesota Living with Heart Failure Questionnaire (MLHFQ) (Turkish version of scale) 21 items rated on six-point Likert scales, representing different degrees of impact of heart failure on Heart Related Quality of Life (HRQoL), from 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst HRQoL), as well as scores for two dimensions, physical (8 items, range 0-40) and emotional (5 items, range 0-25).
Dyspnea | Second day
  It will be evaluated modified Borg Scale. This modified 12-point scale consists (0, 0.5, 1-10) corresponds with increasing shortness of breath. Patients were asked to mark the most appropriate description or number of their shortness of breath at rest and during exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Hanım Eda GÖKTAŞ, MSc, Study Chair — Gazi University; Meral BOŞNAK GÜÇLÜ, PhD, Study Director — Gazi University; Adnan ABACI, PhD, Principal Investigator — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Ankara, Yenimahalle
  - Gazi University Faculty of Health Science Department of Physiotherapy and Rehabilitation, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giannuzzi P, Temporelli PL, Corra U, Tavazzi L; ELVD-CHF Study Group. Antiremodeling effect of long-term exercise training in patients with stable chronic heart failure: results of the Exercise in Left Ventricular Dysfunction and Chronic Heart Failure (ELVD-CHF) Trial. Circulation. 2003 Aug 5;108(5):554-9. doi: 10.1161/01.CIR.0000081780.38477.FA. Epub 2003 Jul 14. PMID 12860904
- [Background] Ades PA, Keteyian SJ, Balady GJ, Houston-Miller N, Kitzman DW, Mancini DM, Rich MW. Cardiac rehabilitation exercise and self-care for chronic heart failure. JACC Heart Fail. 2013 Dec;1(6):540-7. doi: 10.1016/j.jchf.2013.09.002. Epub 2013 Oct 24. PMID 24622007
- [Background] Antunes-Correa LM, Kanamura BY, Melo RC, Nobre TS, Ueno LM, Franco FG, Roveda F, Braga AM, Rondon MU, Brum PC, Barretto AC, Middlekauff HR, Negrao CE. Exercise training improves neurovascular control and functional capacity in heart failure patients regardless of age. Eur J Prev Cardiol. 2012 Aug;19(4):822-9. doi: 10.1177/1741826711414626. Epub 2011 Jun 22. PMID 21697210